CLINICAL TRIAL: NCT05372419
Title: An Open-Label, 24-Week Study to Investigate the Safety and Efficacy of Lebrikizumab in Adult and Adolescent Participants With Moderate-to-Severe Atopic Dermatitis and Skin of Color
Brief Title: A Study of (LY3650150) Lebrikizumab to Assess the Safety and Efficacy of Adult and Adolescent Participants With Moderate-to-Severe Atopic Dermatitis and Skin of Color
Acronym: ADmirable
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18500; J2T-MC-KGBP (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-05-09; First posted 2022-05-12 (Actual); Results first posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Atopic Dermatitis
Keywords: Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — lebrikizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lebrikizumab 250 mg Q2W (Experimental): Participants received a 500 milligram (mg) loading dose of Lebrikizumab subcutaneously (SC) once every 2 weeks (Q2W) at baseline and Week 2, followed by 250 mg SC once Q2W until Week 16.
  Interventions: Drug: Lebrikizumab

INTERVENTIONS:
Drug: Lebrikizumab — Administered SC
  Other Names: LY3650150; DRM06

SUMMARY:
The main purpose of this study is to determine the safety and efficacy lebrikizumab in adolescent and adult participants with moderate-to-severe atopic dermatitis (AD) and skin of color.

ELIGIBILITY:
Inclusion Criteria:

Participants must be ≥12 years of age inclusive, at the time of signing the informed consent/assent.

* Participants who are self-reported race other than White, including but not limited to persons who self-identify as Black or African American, American Indian or Alaska Native, Asian, Native Hawaiian, or Other Pacific Islander.
* Participants who are Fitzpatrick phototype IV-VI
* Participants who have chronic AD that has been present for ≥1 year before screening.
* Have EASI ≥16 at baseline
* Have IGA score ≥3 (Scale of 0 to 4) at baseline
* Have ≥10% body surface area (BSA) of AD involvement at baseline
* Have a history of inadequate response to treatment with topical medications; or determination that topical treatments are otherwise medically inadvisable.
* Adolescents body weight must be ≥40 kg at baseline.
* Are willing and able to comply with all clinic visits and study-related procedures and questionnaires.
* Contraceptive use - Male and/or female

  * Male participants are not required to use any contraception except in compliance with specific local government study requirements.
  * Female participants of child-bearing potential: must agree to remain abstinent (refrain from heterosexual intercourse) or use a highly effective contraceptive method during the treatment period and for at least 18 weeks after the last dose of study drug. Women of non-child-bearing potential (non-WOCBP) may participate without any contraception requirements.

Exclusion Criteria:

* History of human immunodeficiency virus (HIV) infection or positive HIV serology at screening.
* Have a current infection or chronic infection with hepatitis B virus (HBV) at screening, that is, positive for hepatitis B surface antigen (HBsAg) and/or polymerase chain reaction positive for HBV DNA
* Have a current infection with hepatitis C virus (HCV) at screening, that is, positive for HCV RNA
* Have an uncontrolled chronic disease that might require multiple intermittent uses of oral corticosteroids at screening (as defined by the investigator).
* Have uncontrolled asthma that

  * might require bursts of oral or systemic corticosteroids, or
  * required the following due to ≥1 exacerbations within 12 months before baseline

    * systemic (oral and/or parenteral) corticosteroid treatment, or
    * hospitalization for >24 hours.
* Have known liver cirrhosis and/or chronic hepatitis of any etiology.
* Had prior treatment with dupilumab
* Had prior treatment with tralokinumab
* Treatment with topical agents (corticosteroids, calcineurin inhibitors, JAK inhibitors, or phosphodiesterase-4 inhibitors) within 2 weeks prior to baseline.
* Treatment with any of the following agents within 4 weeks prior to the baseline:

  * systemic immunosuppressive/immunomodulating drugs (for example, systemic corticosteroids, cyclosporine, mycophenolate mofetil, IFN-gamma, azathioprine, methotrexate, and other immunosuppressants);
  * small molecules (for example, Janus Kinase (JAK) inhibitors);
  * phototherapy and photochemotherapy for AD.
* History of malignancy, including mycosis fungoides or cutaneous T-cell lymphoma, within 5 years before the screening, except completely treated in situ carcinoma of the cervix of completely treated and resolved non-metastatic squamous or basal cell carcinoma of the skin with no evidence of recurrence in the past 12 weeks.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2025-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (36):
- United States (36):
  - Total Skin and Beauty Dermatology Center, PC, Birmingham, Alabama
  - First OC Dermatology, Fountain Valley, California
  - Center For Dermatology Clinical Research, Inc., Fremont, California
  - Axon Clinical Research, Inglewood, California
  - Avance Clinical Trials Inc, Laguna Niguel, California
  - Dermatology Research Associates, Los Angeles, California
  - Wallace Medical Group, Inc., Los Angeles, California
  - Cura Clinical Research, Palmdale, California
  - University of California Davis (UC Davis) Comprehensive Cancer Center, Sacramento, California
  - Clinical Science Institute, Santa Monica, California
  - Cura Clinical Research, Sherman Oaks, California
  - UConn Health, Farmington, Connecticut
  - Encore Medical Research of Boynton Beach, Boynton Beach, Florida
  - Skin Care Research, Inc, Hollywood, Florida
  - Solutions Through Advanced Research, Jacksonville, Florida
  - Miami Dermatology and Laser Research, Miami, Florida
  - Savin Medical Group, LLC, Miami Lakes, Florida
  - PureSkin Dermatology, Orlando, Florida
  - Skin Care Physicians of Georgia, Macon, Georgia
  - Advanced Medical Research, Sandy Springs, Georgia
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Allcutis Research, Inc., Beverly, Massachusetts
  - Oakland Hills Dermatology, Auburn Hills, Michigan
  - Revival Research Institute - Troy, Troy, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Skin Specialists, P.C, Omaha, Nebraska
  - Sadick Research Group, New York, New York
  - Wilmington Health Family Medicine, Wilmington, North Carolina
  - Dermatology & Laser Center of Charleston, Charleston, South Carolina
  - Arlington Research Center, Inc, Arlington, Texas
  - Clinical Trial Network, Houston, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Complete Dermatology, Sugar Land, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
URL: http://vivli.org/

REFERENCES:
- [Derived] Alexis A, Moiin A, Waibel J, Wallace P, Cohen D, Laquer V, Kwong P, Atwater AR, Schuster C, Proper J, Silk M, Pierce E, Pillai S, Rueda MJ, Moore A; ADmirable Investigators. Efficacy and Safety of Lebrikizumab in Adult and Adolescent Patients with Skin of Color and Moderate-to-Severe Atopic Dermatitis: Results from the Phase IIIb, Open-Label ADmirable Study. Am J Clin Dermatol. 2025 Sep;26(5):803-817. doi: 10.1007/s40257-025-00970-8. Epub 2025 Jul 15. PMID 40665146
- See also: A Study of (LY3650150) Lebrikizumab to Assess the Safety and Efficacy of Adult and Adolescent Participants With Moderate-to-Severe Atopic Dermatitis and Skin of Color — https://trials.lilly.com/en-US/trial/343503

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was designed to be conducted in a 24-week open-label treatment period and a 12-week safety follow-up period. During 24-week treatment period,participants received 500 milligrams (mg) Lebrikizumab subcutaneously (SC) once every 2 weeks (Q2W) at baseline and Week 2, followed by 250 mg Lebrikizumab SC Q2W until Week 16.Responders at Week 16 will receive 250 mg SC once every 4 weeks (Q4W) until Week 24,while inadequate responders will continue with 250 mg Lebrikizumab SC Q2W until Week 24.
Pre-assignment Details: Current results reporting is for the primary outcome, i.e., the open-label treatment period until Week 16. The open-label treatment period Week 24 data and follow-up period data analysis are ongoing and will be presented at the time of reporting the final results, i.e., no later than February 17, 2026.
Period: Overall Study
Arm/Group | Lebrikizumab 250 mg Q2W
Started | 90
Received at Least 1 Confirmed Dose of Study Drug | 90
Completed ("Completed" includes participants who completed the study until Week 16 only. Week 16 to Week 24 data and follow-up period data analysis are ongoing and will be presented at the time of reporting the final results.) | 77
Not Completed | 13
Not completed — Protocol Deviation | 1
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 7

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all enrolled participants according to their planned intervention.
Arm/Group | Lebrikizumab 250 mg Q2W
Number analyzed (Participants) | 90
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.7 (19.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19
  Not Hispanic or Latino | 71
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 4
  Black or African American | 70
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 90

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Eczema Area and Severity Index 75 (≥75% Reduction From Baseline in EASI) at Week 16
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe) at each time point. The EASI75 responder is defined as a ≥ 75% improvement from baseline in the EASI score.
Time Frame: Week 16
Population: ITT population included all enrolled participants according to their planned intervention and had Week 16 EASI 75 data. Observed Cases (OC) analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Lebrikizumab 250 mg Q2W
Number analyzed (Participants) | 78
percentage of participants | 69.2 [60.1 to 77.1]

2. Secondary Outcome: Percentage of Participants Achieving EASI 75 at Week 24
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification, each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe) at each time point. The EASI75 responder is defined as a ≥ 75% improvement from baseline in the EASI score.
  Results for Week 24 data will be presented at the time of reporting the final results.
Time Frame: Week 24
Reporting Status: Not Posted, anticipated posting 2026-02

3. Secondary Outcome: Percentage of Participants With an Investigator's Global Assessment (IGA) Score of 0 or 1 and a Reduction ≥2 Points From Baseline to Week 16
Description: The IGA measures the investigator's global assessment of the participant's overall severity of their AD, based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on the descriptors that best describe the overall appearance of the lesions at a given time point.
Time Frame: Baseline to Week 16
Population: The ITT population included all enrolled participants according to their planned intervention and had a week 16 IGA score of at least 2. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Lebrikizumab 250 mg Q2W
Number analyzed (Participants) | 78
percentage of participants | 44.9 [35.9 to 54.2]

4. Secondary Outcome: Percentage of Participants With an IGA Score of 0 or 1 and a Reduction ≥2 Points From Baseline to Week 24
Description: The IGA measures the investigator's global assessment of the participant's overall severity of their AD, based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on the descriptors that best describe the overall appearance of the lesions at a given time point.
  Results for Week 24 data will be presented at the time of reporting the final results.
Time Frame: Baseline to Week 24
Reporting Status: Not Posted, anticipated posting 2026-02

5. Secondary Outcome: Percentage Change From Baseline in Total EASI Score From Baseline to Week 16
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe) at each time point.
Time Frame: Baseline, Week 16
Population: ITT population included all enrolled participants according to their planned intervention and had Week 16 EASI data. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Lebrikizumab 250 mg Q2W
Number analyzed (Participants) | 78
percentage change | -78.8 (25.33)

6. Secondary Outcome: Percentage Change From Baseline in Total EASI Score From Baseline to Week 24
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe) at each time point.
  Results for Week 24 data will be presented at the time of reporting the final results.
Time Frame: Baseline, Week 24
Reporting Status: Not Posted, anticipated posting 2026-02

7. Secondary Outcome: Change From Baseline in Total EASI Score From Baseline to Week 16
Description: as for outcome 5
Time Frame: Baseline, Week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Lebrikizumab 250 mg Q2W: Participants received a 500 mg loading dose of Lebrikizumab SC once Q2W at baseline and Week 2, followed by 250 mg SC once Q2W until Week 16.
Arm/Group | Lebrikizumab 250 mg Q2W
Number analyzed (Participants) | 78
score on a scale | -20.2 (11.05)

8. Secondary Outcome: Change From Baseline in Total EASI Score From Baseline to Week 24
Description: as for outcome 6
Time Frame: Baseline, Week 24
Reporting Status: Not Posted, anticipated posting 2026-02

9. Secondary Outcome: Percentage of Participants Achieving EASI-90 (≥90% Reduction in EASI Score) From Baseline to Week 16
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe) at each time point. The EASI90 responder is defined as a ≥ 90% improvement from baseline in the EASI score.
Time Frame: Baseline to Week 16
Population: ITT population included all enrolled participants according to their planned intervention and had Week 16 EASI 90 data. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Lebrikizumab 250 mg Q2W
Number analyzed (Participants) | 78
percentage of participants | 44.9 [35.9 to 54.2]

10. Secondary Outcome: Percentage of Participants Achieving EASI-90 From Baseline to Week 24
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe) at each time point. The EASI90 responder is defined as a ≥ 90% improvement from baseline in the EASI score.
  Results for Week 24 data will be presented at the time of reporting the final results.
Time Frame: Baseline to Week 24
Reporting Status: Not Posted, anticipated posting 2026-02

11. Secondary Outcome: Percentage of Participants With a Pruritus Numeric Rating Scale (NRS) of ≥4 Points at Baseline Who Achieve a 4-point Reduction From Baseline to Week 16
Description: Pruritus NRS is an 11-point scale used by participants to rate their worst itch severity over the past 24 hours, with 0 indicating "No itch" and 10 indicating "Worst itch imaginable."
Time Frame: Baseline to Week 16
Population: ITT population included all enrolled participants according to their planned intervention and had week 16 Pruritus NRS score of at least 4. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Lebrikizumab 250 mg Q2W
Number analyzed (Participants) | 62
percentage of participants | 58.1 [47.6 to 67.8]

12. Secondary Outcome: Percentage of Participants With a Pruritus NRS of ≥4 Points at Baseline Who Achieve a 4-point Reduction From Baseline to Week 24
Description: Pruritus NRS is an 11-point scale used by participants to rate their worst itch severity over the past 24 hours, with 0 indicating "No itch" and 10 indicating "Worst itch imaginable."
  Results for Week 24 data will be presented at the time of reporting the final results.
Time Frame: Baseline to Week 24
Reporting Status: Not Posted, anticipated posting 2026-02

13. Secondary Outcome: Percentage of Participants With a Pruritus NRS ≥3 Points at Baseline Who Achieve at Least 3- Point Reduction From Baseline to Week 16
Description: as for outcome 11
Time Frame: Baseline to Week 16
Population: ITT population included all enrolled participants according to their planned intervention and had week 16 Pruritus NRS score of at least 3. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Lebrikizumab 250 mg Q2W
Number analyzed (Participants) | 65
percentage of participants | 66.2 [56.0 to 75.0]

14. Secondary Outcome: Percentage of Participants With a Pruritus NRS ≥3 Points at Baseline Who Achieve at Least 3- Point Reduction From Baseline to Week 24
Description: Pruritus NRS is an 11-point scale used by participants to rate their worst itch severity over the past 24 hours, with 0 indicating "No itch" and 10 indicating "Worst itch imaginable. Assessments were recorded daily by the participant using an electronic diary.
  Results for Week 24 data will be presented at the time of final results reporting.
Time Frame: Baseline to Week 24
Reporting Status: Not Posted, anticipated posting 2026-02

15. Secondary Outcome: Percentage Change in Pruritus NRS Score From Baseline to Week 16
Description: Pruritus NRS is an 11-point scale used by participants to rate their worst itch severity over the past 24 hours, with 0 indicating "No itch" and 10 indicating "Worst itch imaginable." Assessments were recorded daily by the participant using an electronic diary.
Time Frame: Baseline, Week 16
Population: ITT population included all enrolled participants according to their planned intervention and had week 16 pruritus NRS score. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Lebrikizumab 250 mg Q2W
Number analyzed (Participants) | 68
percentage change | -58.3 (36.03)

16. Secondary Outcome: Percentage Change From Baseline in Pruritus NRS Score From Baseline to Week 24
Description: Pruritus NRS is an 11-point scale used by participants to rate their worst itch severity over the past 24 hours, with 0 indicating "No itch" and 10 indicating "Worst itch imaginable." Assessments were recorded daily by the participant using an electronic diary.
  Results for Week 24 data will be presented at the time of reporting the final results.
Time Frame: Baseline, Week 24
Reporting Status: Not Posted, anticipated posting 2026-02

17. Secondary Outcome: Percentage of Participants With a Sleep-Loss Scale Score of ≥2 Points at Baseline Who Achieve a 2-point Reduction From Baseline to Week 16
Description: Sleep loss due to interference of itch will be assessed by the participant. Participants rate their interference of itch on sleep based on a 5-point Likert scale [0 (not at all) to 4 (unable to sleep at all). Higher scores indicated a greater impact and worse outcome. Assessments will be recorded daily by the participant.
Time Frame: Baseline to Week 16
Population: ITT population included all enrolled participants according to their planned intervention and had a baseline Sleep-Loss scale score of at least 2. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Lebrikizumab 250 mg Q2W
Number analyzed (Participants) | 39
percentage of participants | 30.8 [20.2 to 43.8]

18. Secondary Outcome: Percentage of Participants With a Sleep-Loss Scale Score of ≥2 Points at Baseline Who Achieve a 2-point Reduction From Baseline to Week 24
Description: Sleep loss due to interference of itch will be assessed by the participant. Participants rate their interference of itch on sleep based on a 5-point Likert scale [0 (not at all) to 4 (unable to sleep at all). Higher scores indicated a greater impact and worse outcome. Assessments will be recorded daily by the participant.
  Results for Week 24 data will be presented at the time of reporting the final results.
Time Frame: Baseline to Week 24
Reporting Status: Not Posted, anticipated posting 2026-02

19. Secondary Outcome: Percentage Change From Baseline in Sleep-Loss Scale Score From Baseline to Week 16
Description: as for outcome 17
Time Frame: Baseline, Week 16
Population: ITT population included all enrolled participants according to their planned intervention and had week 16 Sleep-Loss scale score. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Lebrikizumab 250 mg Q2W
Number analyzed (Participants) | 63
percentage change | -54.3 (53.52)

20. Secondary Outcome: Percentage Change From Baseline in Sleep-Loss Scale Score From Baseline to Week 24
Description: as for outcome 18
Time Frame: Baseline, Week 24
Reporting Status: Not Posted, anticipated posting 2026-02

21. Secondary Outcome: Percentage of Participants With a Skin Pain NRS of ≥4 Points at Baseline Who Achieve a 4-point Reduction From Baseline to Week 16
Description: The Skin Pain NRS is an 11-point scale used by participants to rate their worst level of skin pain over the past 24 hours, with 0 indicating "no pain" and 10 indicating "worst pain imaginable."
Time Frame: Baseline to Week 16
Population: ITT population included all enrolled participants according to their planned intervention and had week 16 skin pain NRS score of at least 4. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Lebrikizumab 250 mg Q2W
Number analyzed (Participants) | 51
percentage of participants | 58.8 [47.3 to 69.4]

22. Secondary Outcome: Percentage of Participants With a Skin Pain NRS of ≥4 Points at Baseline Who Achieve a 4-point Reduction From Baseline to Week 24
Description: The Skin Pain NRS is an 11-point scale used by participants to rate their worst level of skin pain over the past 24 hours, with 0 indicating "no pain" and 10 indicating "worst pain imaginable."
  Results for Week 24 data will be presented at the time of reporting the final results.
Time Frame: Baseline to Week 24
Reporting Status: Not Posted, anticipated posting 2026-02

23. Secondary Outcome: Change From Baseline inPatient-Oriented Eczema Measure (POEM) From Baseline to Week 16
Description: The POEM is a simple, participant-reported, 7-item scale that assesses disease severity in children and adults. Participants respond to questions about the frequency of 7 symptoms (itching, sleep disturbance, bleeding, weeping/oozing, cracking, flaking, and dryness/roughness) over the past week. Response categories include "No days," "1-2 days," "3-4 days," "5-6 days," and "Every day" with corresponding scores of 0, 1, 2, 3, and 4, respectively The sum of the 7 items gives the total POEM score of 0 (absent disease) to 28 (severe disease). High scores are indicative of more severe disease and poor quality of life.
Time Frame: Baseline, Week 16
Population: ITT population included all enrolled participants according to their planned intervention and had week 16 POEM data. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lebrikizumab 250 mg Q2W
Number analyzed (Participants) | 45
score on a scale | -10.8 (7.51)

24. Secondary Outcome: Change From Baseline in POEM From Baseline to Week 24
Description: The POEM is a simple, participant-reported, 7-item scale that assesses disease severity in children and adults. Participants respond to questions about the frequency of 7 symptoms (itching, sleep disturbance, bleeding, weeping/oozing, cracking, flaking, and dryness/roughness) over the past week. Response categories include "No days," "1-2 days," "3-4 days," "5-6 days," and "Every day" with corresponding scores of 0, 1, 2, 3, and 4, respectively The sum of the 7 items gives the total POEM score of 0 (absent disease) to 28 (severe disease). High scores are indicative of more severe disease and poor quality of life.
  Results for Week 24 data will be presented at the time of reporting the final results.
Time Frame: Baseline, Week 24
Reporting Status: Not Posted, anticipated posting 2026-02

25. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) From Baseline to Week 16
Description: The DLQI questionnaire designed for participants aged >=16 years or more is a 10-item, validated questionnaire used to assess the impact of skin disease on the quality of life of an affected person. The 10 questions cover the following topics: symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment, over the previous week. Response categories include "Not at all," "A little," "A lot," and "Very much," with corresponding scores of 0, 1, 2, and 3 respectively. Questions 3-10 also have an additional response category of "Not relevant" which is scored as "0". Questions are scored from 0 to 3, giving a possible total score range from 0 (no impact of skin disease on quality of life) to 30 (maximum impact on quality of life). A high score is indicative of a poor quality of life.
Time Frame: Baseline, Week 16
Population: The ITT population included all enrolled participants according to their planned intervention and had week 16 DLQI score. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lebrikizumab 250 mg Q2W
Number analyzed (Participants) | 66
score on a scale | -7.4 (6.63)

26. Secondary Outcome: Change From Baseline in DLQI From Baseline to Week 24
Description: The DLQI questionnaire designed for participants aged >=16 years or more is a 10-item, validated questionnaire used to assess the impact of skin disease on the quality of life of an affected person. The 10 questions cover the following topics: symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment, over the previous week. Response categories include "Not at all," "A little," "A lot," and "Very much," with corresponding scores of 0, 1, 2, and 3 respectively. Questions 3-10 also have an additional response category of "Not relevant" which is scored as "0". Questions are scored from 0 to 3, giving a possible total score range from 0 (no impact of skin disease on quality of life) to 30 (maximum impact on quality of life). A high score is indicative of a poor quality of life.
  Results for Week 24 data will be presented at the time of reporting the final results.
Time Frame: Baseline, Week 24
Reporting Status: Not Posted, anticipated posting 2026-02

27. Secondary Outcome: Change From Baseline in Children's Dermatology Life Quality Index (cDLQI) From Baseline to Week 16
Description: The CDLQI questionnaire designed for participants aged <16 years and It consists of 10 items that are grouped into 6 domains: symptoms & feelings, leisure, school or holidays, personal relationships, sleep, & treatment. The scoring of each question is: Very much =3; Quite a lot = 2; Only a little = 1; Not at all = 0. CDLQI total score is calculated by summing all 10 items responses and has a range of 0 to 30 (higher scores are indicative of greater impairment).
Time Frame: Baseline, Week 16
Population: ITT population included all enrolled participants according to their planned intervention and had week 16 CDLQI score. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lebrikizumab 250 mg Q2W
Number analyzed (Participants) | 9
score on a scale | -9.4 (8.50)

28. Secondary Outcome: Change From Baseline in cDLQI From Baseline to Week 24
Description: The CDLQI questionnaire designed for participants aged <16 years and It consists of 10 items that are grouped into 6 domains: symptoms & feelings, leisure, school or holidays, personal relationships, sleep, & treatment. The scoring of each question is: Very much =3; Quite a lot = 2; Only a little = 1; Not at all = 0. CDLQI total score is calculated by summing all 10 items responses and has a range of 0 to 30 (higher scores are indicative of greater impairment).
  Results for Week 24 data will be presented at the time of reporting the final results.
Time Frame: Baseline, Week 24
Reporting Status: Not Posted, anticipated posting 2026-02

29. Secondary Outcome: Percentage of Participants With a DLQI of ≥4 Points at Baseline Who Achieve a ≥4-point Improvement in DLQI From Baseline to Week 16
Description: The DLQI questionnaire for participants aged 16 and above is a 10-item tool used to assess the impact of skin disease on quality of life. The 10 questions cover topics: symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment over the previous week. Response categories include "not at all," "a little," "a lot," and "very much," with corresponding scores of 0, 1, 2, and 3, respectively. Questions 3-10 have an additional response category of "not relevant," which is scored as "0." Questions are scored from 0 to 3. Total score ranges from 0 (no impact) to 30 (maximum impact), with higher scores indicating poorer quality of life.
Time Frame: Baseline to Week 16
Population: ITT population included all enrolled participants according to their planned intervention and had week 16 DLQI score of at least 4. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Lebrikizumab 250 mg Q2W
Number analyzed (Participants) | 60
percentage of participants | 71.7 [61.3 to 80.1]

30. Secondary Outcome: Percentage of Participants With a DLQI of ≥4 Points at Baseline Who Achieve a ≥4-point Improvement in DLQI From Baseline to Week 24
Description: The DLQI questionnaire for participants aged 16 and above is a 10-item tool used to assess the impact of skin disease on quality of life. The 10 questions cover topics: symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment over the previous week. Response categories include "not at all," "a little," "a lot," and "very much," with corresponding scores of 0, 1, 2, and 3, respectively. Questions 3-10 have an additional response category of "not relevant," which is scored as "0." Questions are scored from 0 to 3. Total score ranges from 0 (no impact) to 30 (maximum impact), with higher scores indicating poorer quality of life.
  Results for Week 24 data will be presented at the time of reporting the final results.
Time Frame: Baseline to Week 24
Reporting Status: Not Posted, anticipated posting 2026-02

ADVERSE EVENTS:
Time Frame: Baseline Up to Week 16
Description: All enrolled participants who received at least one confirmed dose of 250 mg lebrikizumab.
  Safety data from the open-label treatment period (Week 24 data) and follow-up period data will be reported during the final results posting, i.e., no later than February 17, 2026.
Arm/Group | Lebrikizumab 250 mg Q2W
All-Cause Mortality (participants affected / at risk) | 0/90
Serious Adverse Events (participants affected / at risk) | 0/90
Other Adverse Events (participants affected / at risk) | 23/90
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lebrikizumab 250 mg Q2W (N=90)
Tachycardia (Cardiac disorders) | 1 (1)
Blepharitis (Eye disorders) | 1 (2)
Dry eye (Eye disorders) | 1 (1)
Diabetic gastroparesis (Gastrointestinal disorders) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1)
Impetigo (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2)
Pustule (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (2)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acanthosis nigricans (Skin and subcutaneous tissue disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-09-29): https://cdn.clinicaltrials.gov/large-docs/19/NCT05372419/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/19/NCT05372419/SAP_001.pdf